CLINICAL TRIAL: NCT02658383
Title: Community-Based Participatory Research: A Tool to Advance Cookstove Interventions
Brief Title: Community-Engaged Research: A Tool to Advance Cookstove Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-3870H; R00ES022269 (NIH)
Record Dates: First submitted 2015-08-24; First posted 2016-01-18 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Blood Pressure; Inflammation; Glycated Hemoglobin (HbA1c)
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cleaner cookstove received after visit 2 (Experimental): This arm receives the cleaner cookstove earlier in the study (after visit 2 which is approximately after 6 months)
  Interventions: Other: Cleaner cookstove received after visit 2
- Cleaner cookstove received after visit 4 (Experimental): This arm receives the cleaner cookstove later in the study (thus acting as a control arm until after visit 4 which is after approximately 1 yr and 6 months)
  Interventions: Other: Cleaner cookstove received after visit 4

INTERVENTIONS:
Other: Cleaner cookstove received after visit 2 — The participants will change from a traditional wood burning cookstove to a cleaner burning (wood) cookstove called the JUSTA (after visit 2).
  Arms: Cleaner cookstove received after visit 2
Other: Cleaner cookstove received after visit 4 — The participants will change from a traditional wood burning cookstove to a cleaner burning (wood) cookstove called the JUSTA (after visit 4).
  Arms: Cleaner cookstove received after visit 4

SUMMARY:
Nearly 3 billion people rely on biomass combustion to meet basic domestic energy needs. Many households use traditional cookstoves to meet these energy needs, which can result in extremely high indoor air pollution concentrations. Indoor air pollution from biomass combustion accounts for an estimated 3.9 million premature deaths per year, representing about 4.8% of the global disease burden. Improved stove designs have the potential to substantially reduce indoor air pollution exposures. However, there are few randomized intervention trials, and previous stove intervention studies have been plagued by low improved stove adoption and sustained use, severely limiting interpretations of these studies. This research proposes to conduct community surveys and in-depth interviews among Honduran cookstove users to gain insight into the complex pathways surrounding barriers to and predictors of sustained improved cookstove adoption (among the target population for the proposed intervention). This information will be used to conduct and enhance a randomized improved cookstove intervention among 300 Honduran families, incorporating qualitative and quantitative measures of cookstove use and measuring pre- to post-intervention changes in pollutant exposures and subclinical indicators of cardiovascular health.

The primary goals are twofold:

* To incorporate community-engaged approaches throughout all aspects of the research
* To maximize sustained stove use (thereby maximizing the health impact of the intervention) to achieve valid exposure-response estimates.

Both objectives utilize innovative strategies to fill knowledge gaps. The research team will build upon previous studies in Latin America that have focused on identifying and validating appropriate field techniques for exposure and health assessments in rural areas of developing countries.

In summary, the proposed project will provide insight regarding barriers/predictors of sustained cookstove adoption, an issue impeding research in this field; assess the relationship between stove use and indicators of cardiovascular health, a substantial and quickly growing disease burden in developing countries; and result in a more comprehensive and valid assessment of the impact of a cookstove intervention.

ELIGIBILITY:
Inclusion Criteria:

* Primary cooks for the household
* Uses a traditional stove
* Latina women (representative of the rural Honduran population, no exclusions based on race/ethnicity)

Exclusion Criteria:

* Non-smoking
* Not pregnant

Ages: 24 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 222 (Actual)
Dates: Start 2015-08; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in Blood pressure | The cleaner burning cookstove will be installed in the homes after 2 visits (after approximately 6 months) and after 4 visits (after approximately 1 yr and 6 months) for half of the population, respectively.
  Intention to treat analyses will incorporate the repeated measures within participants and the change in blood pressure comparing assigned stove type will be the primary outcome of interest. Blood pressure is measured at each of 6 visits spaced approximately 6 months apart over the course of 2.5 years.
Change in glycated hemoglobin (HbA1c) | The cleaner burning cookstove will be installed in the homes after 2 visits (after approximately 6 months) and after 4 visits (after approximately 1 yr and 6 months) for half of the population, respectively.
  Intention to treat analyses will incorporate the repeated measures within participants and the change in HbA1c comparing assigned stove type will be the primary outcome of interest. Blood pressure is measured at each of 6 visits spaced approximately 6 months apart over the course of 2.5 years.
Change in C-reactive protein (CRP) | The cleaner burning cookstove will be installed in the homes after 2 visits (after approximately 6 months) and after 4 visits (after approximately 1 yr and 6 months) for half of the population, respectively.
  Intention to treat analyses will incorporate the repeated measures within participants and the change in CRP comparing assigned stove type will be the primary outcome of interest. Blood pressure is measured at each of 6 visits spaced approximately 6 months apart over the course of 2.5 years.

SECONDARY OUTCOMES:
Change in Inflammation | The cleaner burning cookstove will be installed in the homes after 2 visits (after approximately 6 months) and after 4 visits (after approximately 1 yr and 6 months) for half of the population, respectively.
  Inflammatory markers will be measured in dried blood spots collected at each of 6 visits spaced approximately 6 months apart. Exhaled nitric oxide will also be measured at each visit to assess pulmonary inflammation (in a subset of the population). The lab will analyze the dried blood spots after the completion of the study (not at each 6 month interval); planned inflammatory markers (apart from C-reactive protein, which is a primary outcome) are intracellular adhesion molecule (ICAM-1), Serum amyloid A, and vascular endothelial cell adhesion molecule (VCAM-1)
Change in metabolomics | The cleaner burning cookstove will be installed in the homes after 2 visits (after approximately 6 months) and after 4 visits (after approximately 1 yr and 6 months) for half of the population, respectively.
  The lab will analyze the dried blood spots for untargeted metabolomics after the completion of the study (not at each 6 month interval).
Change in augmentation index and central pulse pressure | The cleaner burning cookstove will be installed in the homes after 2 visits (after approximately 6 months) and after 4 visits (after approximately 1 yr and 6 months) for half of the population, respectively.
  These outcomes will be assessed using the SphygmoCor XCEL.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie L Clark, PhD, Principal Investigator — Colorado State University
Locations (1):
- Field site in Honduras, La Esperanza, Intibucá Department, Honduras

REFERENCES:
- [Background] Young BN, Peel JL, Benka-Coker ML, Rajkumar S, Walker ES, Brook RD, Nelson TL, Volckens J, L'Orange C, Good N, Quinn C, Keller JP, Weller ZD, Africano S, Osorto Pinel AB, Clark ML. Study protocol for a stepped-wedge randomized cookstove intervention in rural Honduras: household air pollution and cardiometabolic health. BMC Public Health. 2019 Jul 8;19(1):903. doi: 10.1186/s12889-019-7214-2. PMID 31286921
- [Result] Young BN, Good N, Peel JL, Benka-Coker ML, Keller JP, Rajkumar S, Walker ES, Volckens J, L'Orange C, Quinn C, Africano S, Osorto Pinel AB, Clark ML. Reduced Black Carbon Concentrations following a Three-Year Stepped-Wedge Randomized Trial of the Wood-Burning Justa Cookstove in Rural Honduras. Environ Sci Technol Lett. 2022 Jun 14;9(6):538-542. doi: 10.1021/acs.estlett.2c00098. Epub 2022 May 4. PMID 38037640
- [Result] Benka-Coker ML, Young BN, Keller JP, Walker ES, Rajkumar S, Volckens J, Good N, Quinn C, L'Orange C, Weller ZD, Africano S, Osorto Pinel AB, Peel JL, Clark ML. Impact of the wood-burning Justa cookstove on fine particulate matter exposure: A stepped-wedge randomized trial in rural Honduras. Sci Total Environ. 2021 May 1;767:144369. doi: 10.1016/j.scitotenv.2020.144369. Epub 2020 Dec 29. PMID 33429278